CLINICAL TRIAL: NCT02517424
Title: Placebo-Controlled, Triple-Blind, Crossover Study of the Safety and Efficacy of Three Different Potencies of Vaporized Cannabis in 42 Participants With Chronic, Treatment-Resistant Posttraumatic Stress Disorder (PTSD)
Brief Title: Evaluating Safety and Efficacy of Cannabis in Participants With Chronic Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tilray (Industry)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CMJP-1
Record Dates: First submitted 2015-07-31; First posted 2015-08-07 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High THC/Low CBD Cannabis (Experimental): Investigational product will be administered via vaporization up to 2 grams per day as needed.
  Interventions: Drug: High THC/Low CBD Cannabis
- High THC/High CBD cannabis (Experimental): Investigational product will be administered via vaporization up to 2 grams per day as needed.
  Interventions: Drug: High THC/High CBD Cannabis
- Low THC/Low CBD cannabis (Placebo Comparator): Product will be administered via vaporization up to 2 grams per day as needed.
  Interventions: Drug: Low THC/Low CBD Cannabis

INTERVENTIONS:
Drug: High THC/Low CBD Cannabis — Dried cannabis
  Arms: High THC/Low CBD Cannabis
Drug: High THC/High CBD Cannabis — Dried cannabis
  Arms: High THC/High CBD cannabis
Drug: Low THC/Low CBD Cannabis — Dried cannabis
  Arms: Low THC/Low CBD cannabis

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of vaporized cannabis in participants with chronic, treatment-resistant posttraumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-5 criteria for chronic PTSD of at least six months duration.
2. Have PTSD of moderate severity as measured by a score of >= 40 on the PCL-5 at the time of baseline assessment.
3. Have treatment resistant PTSD defined as meeting DSM-5 diagnostic criteria for PTSD after failing on, or being unable to tolerate, Health Canada-approved medication or empirically supported psychotherapy for PTSD of adequate dose and duration, as determined on a case-by-case basis by the site investigators.
4. Are at least 18 years old.
5. Are willing to commit to medication dosing and delivery method, to completing evaluation instruments, and to attending all study visits.
6. Agree to use only cannabis provided by study staff until the end of Stage 2 and agree to required cessation periods for the duration of the study.
7. Report no current hazardous cannabis use, as defined by a score of < 11 on the CUDIT-R at time of screening.
8. Abstain from cannabis during the 8-week baseline assessment period as biochemically verified via urine cannabinoid concentrations.
9. Agree to keep all study cannabis stored in a secure location and not to share/distribute cannabis to any other individual.
10. Be stable on medications and/or psychotherapy for PTSD for at least one month prior to study entry.
11. Agree to report any changes in medication or psychotherapy treatment regimen during the study to study staff.
12. If female and of childbearing potential, agree to use an effective form of birth control during study participation.
13. Participants must be proficient in reading English, and must be able to effectively communicate with the investigators and other site personnel.
14. Agree not to participate in any other interventional clinical trials during study participation.
15. Agree not to donate blood from the start of study treatment to 24 hours after the last dose.
16. Agree to allow the collection of his/her gender, race, and occupation to ensure that the study recruits the targeted population.

Exclusion Criteria:

1. Are pregnant or nursing, or of child bearing potential and not practicing an effective means of birth control.
2. Have a history of primary psychotic disorder, bipolar affective disorder, bipolar disorder with psychotic features, depressive disorder with psychotic features, borderline personality disorder, antisocial personality disorder, or positive family history (first degree relative) of psychotic disorder or bipolar affective disorder.
3. Have any allergies to cannabis or contraindication for using cannabis.
4. Are currently taking drugs known to be substrates for CYP 3A4 or CYP 2C19, such as amitriptyline, fentanyl, sufentanil, and alfentanil.
5. Have a diagnosis of obstructive sleep apnea or a score of >3 on the STOP-Bang questionnaire (except in cases where the participant has documented evidence of not having obstructive sleep apnea OR if the participant is compliant on CPAP treatment). Documented evidence consists of a negative result for obstructive sleep apnea on the completion of a formal assessment for apnea.
6. Would present a serious suicide risk as assessed by the investigators, or who are likely to require psychiatric hospitalization during the course of the study.
7. Are not able to give adequate informed consent.
8. Are not able to attend face-to-face visits or plan to move out of the area during the active treatment period.
9. Have a positive urine drug screen for opiates (unless prescribed or contained in an over-the-counter Health Canada approved medication), methamphetamine, cocaine and amphetamines or meet the DSM-5 criteria for substance use disorder (other than caffeine or nicotine) during Stage 1 and 2 of the study.
10. Have signs of ischemia (defined as ST elevation or depression) or significant arrhythmia (defined as atrial fibrillation or flutter, ventricular fibrillation or flutter) on the screening electrocardiogram.
11. Have abnormal hepatic or renal function (abnormal liver function tests or elevated creatinine results on the screening laboratory reports).
12. During the 8-week screening period, are diagnosed with dissociative identity disorder or an eating disorder with active purging, evidence of significant, uncontrolled hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, gastrointestinal, or neurological disease;
13. During the 8-week screening period, meet criteria for cannabis use disorder (4 or more of 11 DSM-5 criteria) and continued cannabis use confirmed by urine testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of Stage 1 in posttraumatic stress disorder symptoms via Clinician Administered PTSD Scale (CAPS) for Diagnostic and Statistical Manual of Mental Disorders (DSM) | 3 weeks

SECONDARY OUTCOMES:
Change in PTSD symptoms during Stage 1 using PTSD Checklist 5 (PCL 5). | 3 weeks
Change in PTSD symptoms during Stage 2 using PCL 5 checklist. | 3 weeks
Change in symptoms of anxiety in Stage 1 via the Inventory of Depression and Anxiety Scale | 3 weeks
Change in symptoms of anxiety in Stage 2 via the Inventory of Depression and Anxiety Scale | 3 weeks
Change in symptoms of depression in Stage 2 via the Inventory of Depression and Anxiety Scale | 3 weeks
Change in psychosocial functioning in Stage 2 via the Inventory of Psychosocial Functioning | 3 weeks
Preference for Stage 1 vs Stage 2 cannabis using the Long-term Follow-up Questionnaire | 34 weeks
Change in PTSD symptoms via CAPS assessment over Stage 1 and 2. | 8 weeks
Change in PTSD symptoms via PCL-5 assessment during abstinence periods. | 2 weeks
Change in sleep quality via actigraphy measures | 10 weeks
Change in sleep quality via Insomnia Severity Index | 8 weeks
Change in sleep quality via Sleep Diary entries | 8 weeks

OTHER OUTCOMES:
Pulse rate following controlled self-administration of investigational product | Day 0
Cannabis withdrawal symptoms | For 2 weeks after administration period
Change in problems associated with cannabis use based on Cannabis Use Disorders Identification Test | 36 weeks
Subjective drug effect via completion of the Drug Effect Questionnaire | For 3 weeks in stage 1 and stage 2, respectively
Presence of suicidal thoughts or behaviors via Columbia Suicide Severity Rating Scale | 36 weeks
Vital signs | 0-10 weeks
Dosing compliance via diary entry and product returns | 0-10 weeks
Abstinence compliance via urine cannabinoid levels | -2 to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zach Walsh, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada